CLINICAL TRIAL: NCT05716477
Title: The Ohio State University Guardant Shield™ Colorectal Cancer Screening Project
Brief Title: Blood Test (Guardant Shield™) for Screening of Colorectal Cancer in Underserved Patients
Status: Completed | Type: Observational
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: Guardant Health, Inc. (Industry)
Responsible Party: Principal Investigator, Electra Paskett, Principal Investigator, Ohio State University Comprehensive Cancer Center
Other Study IDs: OSU-22204; NCI-2023-00078 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2023-01-19; First posted 2023-02-08 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2023-03

CONDITIONS: Colorectal Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Screening (biospecimen collection): Participants undergo blood specimen collection and complete survey on study. Participants may optionally undergo standard of care FIT testing on study.
  Interventions: Procedure: Biospecimen Collection; Other: Survey Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Survey Administration — Complete survey

SUMMARY:
This clinical trial evaluates the use of a blood test (Guardant Shield™) for colorectal cancer screening. Colorectal cancer is the third leading cancer and cause of death in the United States. Screening may help doctors find colorectal cancer early when it is easier to treat yet nearly a third of all people eligible for screening have never had a screening test performed. Currently, doctors use a stool- based test such as the fecal immunochemical test (FIT) and visual tests such as a colonoscopy. Blood based testing such as Guardant Shield™, may provide a quick and effective way to screen patients that are hard to reach or with limited access (underserved).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Recruit women age 45 years and older who are in need of colorectal cancer screening from minority and underserved populations via a community mammography van.

II. Obtain data regarding knowledge, attitudes and beliefs about colorectal cancer screening.

OUTLINE:

Participants undergo blood specimen collection and complete survey on study. Participants may optionally undergo standard of care FIT testing on study.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 45 years of age and older who are in need of colorectal screening
* Do not have a history of cancer
* Able to read and understand English
* Have a provider to receive the results of the test and who will follow-up test results
* Able to provide informed consent

Min Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Recruit women age 45 years and older who are in need of colorectal cancer screening from minority and underserved populations via a community mammography van.
Sampling Method: Non-Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2022-12-23 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Number of patients consented | Up to 2 years
  The number and percentage of patients consented out of those approached to be summarized.
Percentage of patients consented | Up to 2 years
  The number and percentage of patients consented out of those approached to be summarized.
Knowledge about colorectal screening | Up to 2 years
  Summary statistics and data graphics (boxplots, scatterplots, lattice plots) will summarize data about colorectal screening from overall sample and will be correlated with patient demographics using appropriate statistical tests depending on the nature of the data (correlations, t-tests, chi-squared tests, etc.).
Attitudes about colorectal screening | Up to 2 years
  Summary statistics and data graphics (boxplots, scatterplots, lattice plots) will summarize data about colorectal screening from overall sample and will be correlated with patient demographics using appropriate statistical tests depending on the nature of the data (correlations, t-tests, chi-squared tests, etc.).
Beliefs about colorectal screening | Up to 2 years
  Summary statistics and data graphics (boxplots, scatterplots, lattice plots) will summarize data about colorectal screening from overall sample and will be correlated with patient demographics using appropriate statistical tests depending on the nature of the data (correlations, t-tests, chi-squared tests, etc.).

CONTACTS AND LOCATIONS:
Overall Officials: Electra D Paskett, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu